CLINICAL TRIAL: NCT07238777
Title: Relationship of MRI-Based Paraspinal Fatty Degeneration With Bone Mineral Density and Sarcopenia Parameters
Brief Title: MRI-Based Paraspinal Fatty Degeneration and Its Association With BMD and Sarcopenia
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principal Investigator, Beylikduzu State Hospital
Other Study IDs: Beylikdüzüstateh19
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study aims to investigate the relationship between MRI-based paraspinal muscle fatty degeneration, bone mineral density (BMD), and sarcopenia parameters in postmenopausal women. A total of 100 participants aged 60-80 years will be included. Lumbar paraspinal fatty infiltration will be evaluated both qualitatively using the Goutallier classification and quantitatively using ImageJ software to calculate muscle area, fat area, fat ratio, and functional muscle area.

BMD and T-scores of the lumbar spine (L1-L4) and femoral neck will be measured using dual-energy X-ray absorptiometry (DXA). Sarcopenia will be diagnosed based on EWGSOP2 criteria, including muscle mass (assessed by bioelectrical impedance analysis), handgrip strength, and physical performance tests (gait speed, SPPB, TUGT, and 5STS). Sarcopenia-specific quality of life will be assessed using the Sarcopenia Quality of Life Questionnaire (SarQoL-TR).

The study aims to clarify the associations among paraspinal muscle quality, bone health, and sarcopenia, providing a comprehensive understanding of muscle-bone interactions in postmenopausal women. Findings may support the use of paraspinal muscle evaluation as a complementary marker in the management of sarcopenia and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 60-80 years
* Postmenopausal status
* Lumbar MRI and DXA scan performed within the past six months
* Willingness to participate and ability to provide written informed consent

Exclusion Criteria:

* History of lumbar spine surgery (e.g., laminectomy, stabilization)
* Pfirrmann grade ≥4 lumbar disc degeneration on MRI¹³
* Secondary osteoporosis or Paget's disease
* Use of walking aids or mobility restrictions
* Neurological or systemic disorders affecting movement, including:
* Parkinson's disease
* Stroke
* Amyotrophic lateral sclerosis (ALS)
* Central or peripheral vertigo
* Severe immobility or inability to complete performance tests
* Presence of a hip prosthesis

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: postmenopausal women aged 60-80 years
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
MRI-derived paraspinal fat ratio | Baseline
  Evaluation of the association between MRI-derived paraspinal fat ratio and lumbar (L1-L4) and femoral neck BMD values measured by DXA.

SECONDARY OUTCOMES:
Lumbar Bone Mineral Density (BMD) | Baseline
  Lumbar (L1-L4) BMD (g/cm²) measured using dual-energy X-ray absorptiometry (DXA).
Lumbar T-Score | Baseline
  T-scores of L1-L4 vertebrae obtained from DXA scans.
Femoral Neck BMD | Baseline
  BMD (g/cm²) and T-score values of the femoral neck measured by DXA.
Femoral Neck T-Score | Baseline
  BMD (g/cm²) and T-score values of the femoral neck measured by DXA.
Sarcopenia-Specific Quality of Life (SarQoL) Total Score | Baseline
  Quality of life specific to sarcopenia was assessed using the validated Turkish version of the Sarcopenia Quality of Life Questionnaire (SarQoL-TR). The questionnaire consists of 55 items across seven domains: physical and mental health, locomotion, body composition, functionality, activities of daily living, leisure activities, and fears. The total score ranges from 0 to 100, with higher scores indicating better quality of life and lower scores reflecting greater functional limitation and poorer health perception related to sarcopenia.
Goutallier Index | Baseline
  The Goutallier classification was used to visually assess the degree of fatty degeneration in the lumbar paraspinal muscles (L1-L4) on axial MRI images. Each level was graded from 0 to 4, where Grade 0 indicates normal muscle without fat, and Grade 4 represents fat content greater than muscle tissue (>50%). Higher grades indicate greater fatty infiltration and poorer muscle quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)